CLINICAL TRIAL: NCT05495503
Title: Evaluation of the Tolerance of Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Post-inflamamatory Hyperpigmentation (PIH).
Brief Title: Tolerance of Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Post-inflamamatory Hyperpigmentation (PIH).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cryonove Pharma (Industry)
Collaborators: Dermatech (Industry); CEISO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CS5_2
Record Dates: First submitted 2022-08-04; First posted 2022-08-10 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Post-inflammatory Hyperpigmentation
Keywords: Cryotherapy; Hyperpigmentation; Skin Diseases
MeSH Terms: conditions — Hyperpigmentation; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prototype (814A-v1) (Experimental): Application of the prototype (814A-v1) at D0 and D7.
  Interventions: Device: Prototype (814A-v1)
- Prototype (814B-v1) (Experimental): Application of the prototype (814B-v1) at D0 and D7.
  Interventions: Device: Prototype (814B-v1)
- Prototype (814C-v1) (Experimental): Application of the prototype (814C-v1) at D0 and D7.
  Interventions: Device: Prototype (814C-v1)
- Prototype (814D-v1) (Experimental): Application of the prototype (814D-v1) at D0 and D7.
  Interventions: Device: Prototype (814D-v1)

INTERVENTIONS:
Device: Prototype (814A-v1) — Application on PIH located on the dorsal area (2 treatments during the study).
  Arms: Prototype (814A-v1)
Device: Prototype (814B-v1) — Application on PIH located on the dorsal area (2 treatments during the study).
  Arms: Prototype (814B-v1)
Device: Prototype (814C-v1) — Application on PIH located on the dorsal area (2 treatments during the study).
  Arms: Prototype (814C-v1)
Device: Prototype (814D-v1) — Application on PIH located on the dorsal area (2 treatments during the study).
  Arms: Prototype (814D-v1)

SUMMARY:
CS5_2 study aims to evaluate the tolerance of 4 different conditions of cryotherapy treatments applied on dorsal post-inflammatory hyperpigmentation (PIH) spots.

This study is a proof of concept, designed to be interventional, monocentric, randomized and double blind.

The study will evaluate 4 prototypes : (814A-v1), (814B-v1), (814C-v1) and (814D-v1).

DETAILED DESCRIPTION:
Background:

Hyperpigmentation is a problem in all skin types. Safe depigmentation is a challenge. Cryotherapy with liquid nitrogen at -70 °C has been used in the treatment of solar skin lesions for many years but causes considerable damage.

Difluoroethane sprays (CRYONOVE) induce skin temperatures from -5 to -15 °C which ablates melanocytes but leaves the other skin cells viable, causing less discomfort and damage. The prototype sprays in this proof of concept study have been proven safe and effective in the treatment of hyperpigmentation (solar lentigines) in Fitzpatrick skin types (FST) I to IV. Although lentigines are uncommon in darker phototypes, hyperpigmentation (PIH and melasma) is a major issue, thus this study seeks to assess the tolerance (acceptability) of the approach in hyperpigmented unexposed dorsal skin.

Following the side effects occurring after conventional cryotherapy application, the sponsor has selected other sequences of a specific cryogenic spray which has been used effectively and safely for lentigos treatment in Fitzpatrick Phototypes I to IV, with benefit for the consumers without any adverse safety outcomes. There is therefore a need to test the devices on darker skin types (Fitzpatrick V and VI), which also encounter hyperpigmentation challenges.

Design:

In this proof of concept study, the sponsor aims to evaluate the tolerance of 4 prototypes of cryogenic spray.

Intervention:

The prototypes are (814A-v1), (814B-v1), (814C-v1) and (814D-v1) and will be applied on PIH located on the dorsal area. Each treatment corresponds to a specific sequence of a cryogenic spray.

12 subjects will be includes to reach at least 48 brown spots treated. The PIH spots must be between ≥ 3 mm to ≤ 6 mm in diameter.

Each spot will be treated by one of a defined prototype (always the same prototype on the same spot all along the study) and will be treated twice during the study with a 15-day interval between each treatment. At D0, D14 for all the prototypes (814A-v1), (814B-v1), (814C-v1) and (814D-v1).

The follow up visits will be programmed at D7, D21, D28 and D56 for the end visit.

In total this study extends over 8 weeks and involves seven visits (D<0 (inclusion visit), D0,D7, D14, D21, D28 and D56).

Prior to any study device application, the dermatologist will assess the adverse events and will decide if the period between the two applications should be extended or not. The dermatologist will verify that the skin has not been treated by cosmetic products (no presence of cream that could interfere with the treatment) and is dry.

An operator previously trained by the dermatologist will apply the study device to the patient's spots.

Subjects will be lying on their abdomen to make application more stable, and the treatment will be administered with device.

ELIGIBILITY:
Inclusion Criteria:

* Female or male.
* African ethnicity
* Ages 18 to 65.
* Phototype V and VI according to Fitzpatrick scale
* Featuring brown spots (PIH) on the back ≥ 3 mm to ≤ 6 mm in diameter (at least 4 spots per subject).
* Agreeing not to be exposed to the sun (or artificial UV) during the study.
* Informed, having undergone a general clinical examination attesting to his ability to participate in the study.
* Having given written consent for participation in the study.
* No suspicion of carcinoma after investigation by a Dermatologist.

Exclusion Criteria:

* Having performed cosmetic treatments (exfoliants, scrubs or self-tanners, UV ...) in the month before the start of the study, at the level of the back.
* Having applied a depilatory or exfoliating product in the month prior to the start of the study, at the level of the back.
* Having performed cosmetic treatments in a dermatologist (laser, Intense Pulsed Light (IPL), peeling, creams, cryotherapy ...), at the level of the back in the last 6 months.
* With dermatosis, autoimmune disease, systemic, chronic or acute disease, or any other pathology that may interfere with treatment or influence the results of the study (people with diabetes or circulatory problems, allergic to cold, Raynaud's syndrome...).
* Receiving treatment by general or local (dermo corticoids, corticosteroids, diuretics, anti-coagulants ...) likely to interfere with the evaluation of the parameter studied.
* Participating in another study or being excluded from a previous study.
* Unable to follow the requirements of the protocol.
* Vulnerable: whose ability or freedom to give or refuse consent is limited.
* Major protected by law (tutorship, curatorship, safeguarding justice...).
* People unable to read and write English language.
* Unable to be contacted urgently over the phone.
* Been on any other medication which may affect the outcome of the study or affect the skin condition in some way.
* Having ever undergone chemotherapy or other radiation treatment or received any prescription medication or medical treatment understood by them to affect the skin condition.
* Having any skin condition otherwise unsuitable for treatment in the opinion of the Investigator or clinician.

For female subjects:

* Pregnant woman (or wishing to be pregnant during study) or while breastfeeding.
* A woman, who does not use effective methods of contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline skin hyperpigmentation | Day 0, Day 7, Day 14, Day 21, Day 28 and Day 56
  Clinical evaluation of outcomes on each selected and treated spot will be performed by a Dermatologist by scoring with standardized position and lighting at each visit and before each treatment.
  The evaluation will be performed visually on the selected spots. A scale in 6 points (0 to 5) will be used : 0=Clear of hyperpigmentation; 1= Almost clear of hyperpigmentation; 2=mild, but noticeable hyperpigmentation; 3=moderate hyperpigmentation (medium brown in quality); 4=severe hyperpigmentation (dark brown in quality); 5= very severe hyperpigmentation (very dark brown, almost black in quality).
Change from baseline skin hypopigmentation | Day 0, Day 7, Day 14, Day 21, Day 28 and Day 56
  Clinical evaluation of outcomes on each selected and treated spot will be performed by a Dermatologist by scoring with standardized position and lighting at each visit and before each treatment.
  The evaluation will be performed visually on the selected spots. A scale in 5 points will be used (0 to 4): 0=no hypopigmented lesion; 1= very slight area of hypopigmentation of very small size and very slightly fairer than the surrounding skin; 2= slight area of hypopigmentation of small size and slightly fairer than the surrounding skin; 3= moderate : area of hypopigmentation of moderate size and much fairer than the surrounding skin; 4= severe : area of hypopigmentation of large size and much fairer than the surrounding skin
Change from baseline skin appearance | Day 0, Day 7, Day 14, Day 21, Day 28 and Day 56
  Clinical evaluation of outcomes on each selected and treated spot will be performed by a Dermatologist by scoring with standardized position and lighting at each visit and before each treatment.
  The evaluation will be performed visually on the selected spots and surrounded spotless skin area around the spot skin to assess erythema, oedema blister, bubble, scars, micro-bruise, hematoma, dryness,desquamation, fissures/cracks, roughness,crust.
  A scale in 5 points (0 to 4) will be used : 0=none; 1=very mild; 2=mild; 3=moderate; 4=severe.
Change from baseline skin sensation | Day 0, Day 7, Day 14, Day 21, Day 28 and Day 56
  Clinical evaluation of outcomes on each selected and treated spot will be performed by a Dermatologist by scoring with standardized position and lighting at each visit and before each treatment.
  The evaluation will be performed visually on the selected spots and around the spot skin to assess tightness, stinging, itching, warm and burning sensation.
  A scale in 5 points (0 to 4) will be used : 0=none; 1=very mild; 2=mild; 3=moderate; 4=severe.
Self-assesment of pain | Day 0
  The pain of the treatment will be assessed by the Visual Analogue Scale (VAS) at time T0 on the treated area.
  The pain assessed is that felt during the application of the devices. It will be collected from the patient within 5 minutes of application.
  The VAS is made up of a 10-centimeter line anchored by two ends of the pain. One end is the "maximum pain imaginable". The other end is "no pain."
Change from baseline spots visibility | Day 0, Day 7, Day 14, Day 21, Day 28 and Day 56
  Standardized photographs will be taken using a Dermatoscope C-Cube® (PIXIENCE). The capture will be taken on the previously selected spot (and spotless surrounding each spot in the same acquisition) and a spotless area (one on back and far from PIH spot).
  Acquisition will be performed at Day0/time 0 (before treatment) and at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Beverley Summers, Principal Investigator — beverley.summers@smu.ac.za
Locations (1):
- Photobiology Laboratory, Sefako Makgatho Health Sciences University, Pretoria, Gauteng, South Africa